CLINICAL TRIAL: NCT02113540
Title: Atorvastatin and Prevention of Contrast Induced Nephropathy Following Coronary Angiography
Brief Title: Assessment of the Effect of Atorvastatin on Prevention of CIN in Patients Undergoing Coronary Angiography
Acronym: CIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, peyman bidram, Dr peyman bidram, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Grant number: 392172
Record Dates: First submitted 2014-04-05; First posted 2014-04-14 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Contrast Induced Nephropathy
Keywords: coronary angiography; chronic stable angina; CIN
MeSH Terms: conditions — Angina, Stable | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- placebo group (Placebo Comparator): taking atorvastatin like placebo 12 hours before the procedure
- long term statin group (No Intervention): taking atorvastatin for a long time before entering the study (their routine treatment)
- preoperation statin group (Experimental): taking atorvastatin 12 hours before the procedure
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin
  Arms: preoperation statin group

SUMMARY:
As the effect of statin use before the angiography to prevent contrast induced nephropathy (CIN) is not well-known, the aim of the current study is to assess the effect of atorvastatin on prevention of CIN in patients undergoing coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* having chronic stable angina who were referred for coronary angiography
* non-pregnant female subjects
* no history of diabetes mellitus
* no history of renal failure
* no history of single kidney
* no history of cardiogenic shock
* no history of unstable angina
* no history of myocardial infarction
* no history of hypersensitivity to statins
* no history of previous intravascular contrast injection during one month before admission

Exclusion Criteria:

* glomerular filtration rate (GFR) <60
* cardiogenic shock

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2012-01; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Contrast induced nephropathy (CIN) incidence | 48 hours after the procedure
  CIN is determined as an increase in post-procedural serum creatinine of > 0.5 mg/dl or > 25% from baseline in the absence of any other causes

SECONDARY OUTCOMES:
serum creatinine (Cr) level | 48 hours after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan, Isfahan, Iran